CLINICAL TRIAL: NCT01922843
Title: A Phase 2B, Double-blind, Randomized, Placebo-controlled, Proof-of-concept Study of an Oral Vitamin D Compound (DP001) in Secondary Hyperparathyroidism in Patients on Hemodialysis
Brief Title: A Phase 2 Study of an Oral Vitamin D Compound (DP001) in Secondary Hyperparathyroidism in Patients on Hemodialysis
Acronym: 2MD-7H-2B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Deltanoid Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2MD-7H-2B
Record Dates: First submitted 2013-08-12; First posted 2013-08-14 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Hyperparathyroidism, Secondary; Kidney Failure, Chronic
Keywords: Hemodialysis
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DP001 (Experimental): DP001 softgel capsules, 440 ng taken orally three times weekly after dialysis for 12 weeks
  Interventions: Drug: DP001 softgel capsules
- Placebo (Placebo Comparator): Placebo softgel capsules, taken orally three times weekly after dialysis for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DP001 softgel capsules
  Other Names: 2-methylene-19-nor-20S-1α,25-(OH)2D3; PF-00217763; 2MD
  Arms: DP001
Drug: Placebo
  Other Names: Placebo soft gel capsules
  Arms: Placebo

SUMMARY:
The goal of this study is to test a new vitamin D compound for its ability to reduce parathyroid hormone levels in patients who are on hemodialysis.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study of the vitamin D analog 2-methylene-19-nor-20S-1α,25-dihydroxyvitamin D3 (DP001) in patients with end-stage renal disease (ESRD). The effect of 12 weeks of oral administration of DP001 on serum parathyroid hormone (PTH) levels will be evaluated in ESRD patients who have secondary hyperparathyroidism.

ELIGIBILITY:
Inclusion Criteria:

* Men and non-pregnant women ≥18 years of age
* Patient is diagnosed with ESRD and must be on hemodialysis 3 times per week for at least 3 months prior to Screening Phase
* Patient is currently being treated with pharmaceutical vitamin D for the treatment of secondary hyperparathyroidism
* Serum iPTH value ≤500 pg/mL at first screening visit
* Total serum calcium (corrected for albumin) ≤10.5 mg/dL at first screening visit
* Serum phosphorus ≤7.0 mg/dL at first screening visit

Exclusion Criteria:

* Currently taking any of the following: drugs affecting vitamin D metabolism, digitalis, glucocorticoids, cyclosporine or other immunosuppressants, aluminum-based phosphate binders
* A daily intake >4000 IU vitamin D (D3 + D2)
* Any investigational drug use within 10 half-lives of the drug (or within the previous 30 days if the half-life of the drug is unknown)
* History of any of the following: ventricular dysrhythmias, severe congestive heart failure, angina pectoris, myocardial infarction, coronary angioplasty, coronary artery bypass grafting, multiple myeloma, calciphylaxis, active malignancy, end-stage liver disease, active infections, clinically significant renal/urinary tract stones, sarcoidosis, tuberculosis, parathyroidectomy
* Major surgery within the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2013-09; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
The proportion of patients who achieve two consecutive > or = 30% decreases from his/her baseline serum iPTH level | 12 weeks, with weekly iPTH measurements

SECONDARY OUTCOMES:
Mean percentage change in serum iPTH | Baseline to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Thadhani, MD, Study Chair — Massachusetts General Hospital
Locations (14):
- United States (14):
  - Phoenix, Arizona
  - Tucson, Arizona
  - Washington D.C., District of Columbia
  - Evanston, Illinois
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Great Neck, New York
  - Ridgewood, New York
  - Charlotte, North Carolina
  - Cincinnati, Ohio
  - Nashville, Tennessee
  - Fort Worth, Texas
  - Grand Prairie, Texas
  - San Antonio, Texas

REFERENCES:
- [Derived] Thadhani R, Zella JB, Knutson DC, Blaser WJ, Plum LA, Clagett-Dame M, Buck RD, DeLuca HF. 2MD (DP001), a Single Agent in the Management of Hemodialysis Patients: A Randomized Trial. Am J Nephrol. 2017;45(1):40-48. doi: 10.1159/000452680. Epub 2016 Nov 24. PMID 27880946